CLINICAL TRIAL: NCT05392725
Title: Epidemiological Study on Malignancy Complicated With Renal Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Lulin Min, Attending, RenJi Hospital
Other Study IDs: KY2021-253-B
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal renal function group: Observe survival time
- Renal dysfunction group: Observe survival time

SUMMARY:
The epidemiological study of tumor complicated with kidney disease can clarify the prevalence and risk factors of renal injury when malignant tumor is diagnosed, and understand the impact of malignant tumor complicated with renal injury on survival time. This study will bring enlightenment to clinicians, discover high-risk factors in time, and try to avoid renal damage factors in diagnosis and treatment. Early diagnosis and early treatment can partially terminate the progress of renal injury, avoid the suspension of treatment due to renal reasons, and avoid the occurrence of end-stage renal failure (ESRD).

DETAILED DESCRIPTION:
1. To determine the prevalence of malignant tumor complicated with renal injury and analyze the related risk factors.
2. To compare the survival time of malignant tumor with or without renal injury

ELIGIBILITY:
Inclusion Criteria:

* Malignancy confirmed by pathology.
* Between 18-80 years old, regardless of gender; Patients initially diagnosed with malignant tumors in our hospital from July 2017 to June 2021; Waiver of informed consent.

Exclusion Criteria:

* Patients with benign tumor diagnosed by pathology; The patient refused to participate; Patients judged by other researchers as unsuitable for inclusion in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients initially diagnosed with malignancy in Shanghai Renji Hospital from July 2017 to June 2021
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
survival | 3 years
  survival time

IPD SHARING:
Plan to Share IPD: No